CLINICAL TRIAL: NCT07292064
Title: Investigation of Type D Personality, Somatization Disorder and Perceived Social Support in Patients With Temporomandibular Joint Disorders
Brief Title: Type D Personality, Somatization and Perceived Social Support in Temporomandibular Joint Disorders
Status: Completed | Type: Observational
Sponsor: Gulseren Demir Karakilic (Other)
Collaborators: Bozok University (Other); Gaziantep City Hospital (Other)
Responsible Party: Sponsor-Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Other Study IDs: 124/2025
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Disorders; Somatization Disorder; Type D Personality; Perceived Social Support
Keywords: Temporomandibular Joint Pain; Psychosocial Factors; Personality Traits; Social Inhibition; Negative Affectivity; Mandibular Function; Anxiety and Depression; Biopsychosocial Model
MeSH Terms: conditions — Temporomandibular Joint Disorders; Somatoform Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Temporomandibular Joint Disorder Group: Adults aged 18-65 years who were clinically diagnosed with temporomandibular joint disorders at the Otorhinolaryngology outpatient clinic of Gaziantep City Hospital. Participants completed questionnaires evaluating mandibular function, anxiety, depression, personality traits, somatization, and perceived social support. No medical or pharmacological intervention was applied.
- Healthy Control Group: Healthy adults aged 18-65 years with no diagnosis or symptoms of temporomandibular joint disorders. The control participants were matched to the patient group by age and gender and completed the same psychological and functional assessment questionnaires.

SUMMARY:
This study aimed to investigate the relationship between Type D personality traits, somatization disorder, and perceived social support in individuals diagnosed with temporomandibular joint disorders. Temporomandibular joint disorders are musculoskeletal and neuromuscular conditions that affect the jaw joint, chewing muscles, and related structures, leading to pain and functional difficulties. Psychological and social factors, such as personality traits and emotional distress, have been shown to influence the development and persistence of these disorders.

The research was conducted as a prospective cross-sectional study between February and June 2025 in Gaziantep City Hospital. Adult participants between 18 and 65 years of age who were diagnosed with temporomandibular joint disorders were compared with healthy individuals of similar age and gender. Participants completed validated questionnaires that assessed mandibular function, anxiety and depression symptoms, Type D personality traits, somatization tendencies, and levels of perceived social support. The purpose of this study was to provide a more comprehensive understanding of the psychological and social dimensions that may contribute to the onset and course of temporomandibular joint disorders.

DETAILED DESCRIPTION:
This research was designed as a prospective cross-sectional study conducted between February 2025 and June 2025 in the Otorhinolaryngology outpatient clinic of Gaziantep City Hospital, Turkey. The study included two groups: patients diagnosed with temporomandibular joint disorders and healthy control participants matched for age and gender. All participants were between 18 and 65 years of age, literate, cognitively intact, and voluntarily agreed to participate. Ethical approval was granted by the institutional ethics committee, and written informed consent was obtained from all individuals before enrollment.

Data collection involved face-to-face interviews using standardized self-report questionnaires. The following instruments were used:

1. **Mandibular Function Impairment Questionnaire:** This instrument includes 17 questions that evaluate functional problems of the jaw during daily activities. Each question is scored on a five-point scale, and higher total scores indicate greater impairment in jaw function.
2. **Hospital Anxiety and Depression Scale:** This tool consists of 14 questions that measure symptoms of anxiety and depression. It has two parts, each containing seven questions. Each section produces a total score between zero and twenty-one, where higher values represent greater symptom severity.
3. **Type D Personality Scale:** This scale contains fourteen statements divided into two categories: negative emotions and social inhibition. Each statement is rated on a five-point scale from zero to four. A score of ten or more on both categories indicates the presence of Type D personality traits.
4. **Somatization Scale:** This questionnaire includes thirty-three true or false statements that identify the presence of unexplained physical symptoms. Some statements are reverse coded. Higher total scores show more frequent or severe somatic complaints.
5. **Multidimensional Scale of Perceived Social Support:** This twelve-question scale measures perceived emotional and practical support from three sources: family, friends, and a significant other. Each item is rated on a seven-point scale. Higher scores represent stronger perceived social support.

In addition to these scales, sociodemographic data such as age, sex, marital status, education, occupation, and income were recorded. Exclusion criteria included the presence of severe psychiatric disorders, neurological disease, or cognitive impairment that could interfere with understanding or completing the questionnaires.

All collected data were analyzed using appropriate statistical methods. Distribution normality was assessed, and comparisons between the two groups were performed using suitable parametric or non-parametric tests. Associations among the measured psychological and functional parameters were examined through correlation analyses.

The objective of this study was to identify potential associations between Type D personality, somatization, and perceived social support in individuals with temporomandibular joint disorders. By evaluating these interrelated psychological and social variables, the study sought to emphasize the importance of a holistic and multidisciplinary approach in understanding and managing temporomandibular joint disorders.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years

Ability to read and write

Cognitively intact

Patients diagnosed with temporomandibular joint disorders or healthy volunteers

Exclusion Criteria:

Younger than 18 years or older than 65 years

Illiteracy

Cognitive impairment

Not meeting the specified inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 65 years who were diagnosed with temporomandibular joint disorders and presented to the Otorhinolaryngology outpatient clinic at Gaziantep City Hospital. In addition, age- and sex-matched healthy volunteers without temporomandibular joint disorders were included as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Type D Personality Traits | At the time of study enrollment.
  The primary outcome of this study was the evaluation of Type D personality traits in individuals with temporomandibular joint disorders compared to healthy controls. Type D personality was assessed with a fourteen-item scale measuring two main dimensions: negative emotions and social inhibition. Each item is scored from zero to four. A score of ten or more in both dimensions indicates the presence of Type D personality traits. The Turkish version of the scale has been validated and shown to be reliable. Higher total scores indicate stronger negative emotional responses and greater social inhibition.
the Somatization Scale | At the time of study enrollment.
  Somatic symptom severity was measured using a thirty-three-item true or false questionnaire. Seventeen items are reverse-coded to control for response bias. One point is given for each correct standard response and for incorrect responses to reverse-coded items. The total score ranges from zero to thirty-three, with higher scores reflecting more pronounced somatization tendencies. The Turkish version of this instrument has demonstrated reliability and construct validity in previous psychometric evaluations.
the Multidimensional Scale of Perceived Social Support | At the time of study enrollment.
  Perceived emotional and practical support was evaluated using a twelve-item questionnaire measuring three main sources of support: family, friends, and a significant other. Each statement is rated on a seven-point scale ranging from one (very strongly disagree) to seven (very strongly agree). Subscale scores range from four to twenty-eight, and total scores range from twelve to eighty-four. Higher scores indicate greater perceived social support. The Turkish version of this scale has been shown to have high reliability and validity

SECONDARY OUTCOMES:
the Hospital Anxiety and Depression Scale | At the time of study enrollment
  Symptoms of anxiety and depression were evaluated using a fourteen-item self-report scale consisting of two subscales, each containing seven items. Each question is scored from zero to three, resulting in subscale scores ranging from zero to twenty-one. Higher scores indicate greater symptom severity. This tool has been validated in Turkish and is widely used to identify possible mood and anxiety symptoms in clinical and research settings.
the Mandibular Function Impairment Questionnaire | At the time of study enrollment.
  Jaw function and movement limitations were evaluated using a seventeen-item questionnaire assessing the degree of difficulty in performing daily activities involving mandibular movement. Each item is rated on a five-point scale from zero (no difficulty) to four (very severe difficulty). The total score ranges from zero to sixty-eight, with higher scores indicating greater functional impairment of the jaw. The Turkish adaptation of this scale has demonstrated strong reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Gülseren Demir Karakılıç, Assistant Professor, Principal Investigator — Yozgat Bozok University
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and analyzed during the current study will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The individual participant data and supporting documents will be available beginning six months after publication of the main results and will remain available for a minimum of five years.
Access Criteria: Individual participant data and supporting documents will be accessible to qualified researchers upon submission of a reasonable request to the corresponding author. Requests should include a methodologically sound research proposal and a commitment to use the data only for research purposes. Data will be shared in de-identified form to protect participant confidentiality.
URL: https://hastane.bozok.edu.tr/

REFERENCES:
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Eker, D., Cok boyutlu algilanan sosyal destek olceginin gozden gecirilmis formunun faktor yapisi, gecerlik ve guvenirligi. Turk Psikiyatri Dergisi, 2001. 12: p. 17-25.
- [Background] Dülgerler, Ş., İlköğretim okulu öğretmenlerinde somatizasyon ölçeğinin geçerlik ve güvenirlik çalışması. Unpublished master dissertation). Ege University, İzmir, 2000.
- [Background] Öncü, E. and S.K. Vayısoğlu, D tipi kişilik ölçeğinin Türk toplumunda geçerlilik ve güvenirlilik çalışması. Ankara Medical Journal, 2018. 18(4): p. 646-656.
- [Background] Denollet J. DS14: standard assessment of negative affectivity, social inhibition, and Type D personality. Psychosom Med. 2005 Jan-Feb;67(1):89-97. doi: 10.1097/01.psy.0000149256.81953.49. PMID 15673629
- [Background] Aydemir, Ö., et al., Validity and reliability of Turkish version of hospital anxiety and depression scale. Turk Psikiyatri Derg, 1997. 8(4): p. 280-7.
- [Background] Kılınç, H.E., et al., Further Validity and Reliability of Turkish Version of the Mandibular Functional Impairment Questionnaire in Patients with Temporomandibular Dysfunction. Journal of Basic and Clinical Health Sciences, 2022. 7(1): p. 214-222.